CLINICAL TRIAL: NCT06513117
Title: LIving BEtteR With asThma studY: A Multimodal Intervention to Address Multimorbidity in Difficult Asthma
Brief Title: LIving BEtteR With asThma studY:: A Multimodal Intervention to Address Multimorbidity in Difficult Asthma
Acronym: LIBERTY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM RSP 0002
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Asthma; Multi Morbidity
Keywords: exercise; behaviour change; multimorbidity; asthma
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pilot single arm trial of a structured responsive exercise program and psychological/behavioural support.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Intervention (Exercise, breathing retraining nutritional and behaviour change support) (Experimental): Participants with difficult asthma and multimorbidity (more than 2 additional long term health conditions alongside asthma) will be invited to take part in the study. Participants will undertake in a 6-month/ 24 week supervised multimodal health improvement programme (combining exercise training, behavioural change support, breathing retraining and dietary and emotional self-management support. This programme will run alongside usual treatment.
  Participants will be asked to undergo some additional exercise-based tests, activity monitoring, assessment of nutritional wellbeing and complete some questionnaires before, after and during the intervention, with a total of 3 face to face study visits and 2 virtual visits at University Hospital Southampton.
  Interventions: Behavioral: Behaviour change; Behavioral: Dietary support; Behavioral: Breathing pattern retraining; Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Behaviour change — healthy conversations to support behaviour change
  Other Names: healthy conversations
Behavioral: Dietary support — Guidance on healthy eating
Behavioral: Breathing pattern retraining — guidance on breathing pattern in exercise
Behavioral: Exercise training — Exercise intervention prescribed to participant fitness level

SUMMARY:
Multimorbidity is a significant issue for many patients with difficult asthma. With patients, we have co-designed a multimodal intervention comprising prescribed exercise, dietary support, breathing pattern retraining and behaviour change to target multimorbidity in difficult asthma

DETAILED DESCRIPTION:
Multimorbidity (living with more than 2 additional health conditions) is very common for patients with Difficult Asthma, and has an impact on symptom burden and exacerbation frequency. The investigators want to find out if a personalised intervention (i.e. exercise training, behavioural change support, breathing retraining and dietary and emotional self-management support) to address mutimorbidity is feasible and tolerable and can improve asthma symptoms in difficult asthma. The investigators also want to find out if this intervention continues to benefit patients and help them to continue lifestyle changes after the intervention has finished.

The aim of this exercise training will be to improve fitness. The investigators believe that increases in physical fitness will improve symptom burden through reductions in inflammation and improved resilience. The aim of the dietary and emotional self-management support is to help participants develop their own solutions for healthy eating and keeping emotionally well. The aim of the behavioural change programme is to help participants continue these lifestyle changes post intervention and manage the challenges of living with difficult asthma alongside other multiple health conditions.

This is a pilot study, so all participants will receive the intervention.

Participants with difficult asthma and multimorbidity (more than 2 additional long term health conditions alongside asthma) will be invited to take part in the study. Participants will undertake in a 6-month/ 24 week supervised multimodal health improvement programme (combining exercise training, behavioural change support, breathing retraining and dietary and emotional self-management support. This programme will run alongside their treatment. The programme will be delivered by highly trained Health Guides, who are trained exercise professionals and have received additional training including how to support people to change their behaviour to be able to look after their own physical and emotional wellbeing by themselves in the long run. During the first 12 weeks, participants will take part in 2 community gym based sessions and 1 home based exercise session every week, all supervised by the Health Guide (in person in the gym and through a video or telephone call at home). For weeks 12-24, they will complete 1 community gym based session and 1 virtual/home based session, supervised by the Health Guide, and 1 session on their own. The sessions with the Health Guide will consist of:

* exercise programme, tailored to individual needs and abilities.
* breathing pattern guidance to regulate breathing pattern during exercise.
* conversations with the Health Guide to support changing diet if needed or keeping up with a healthy diet if they already eat healthily.
* conversations with Health Guide to support in becoming confident to exercise on their own and finding own ways of keeping physically active in the long run.
* conversations about emotional wellbeing and how to look after emotional health Participants will be asked to undergo some additional exercise-based tests, activity monitoring, assessment of nutritional wellbeing and complete some questionnaires before, after and during the intervention, with a total of 3 face to face study visits and 2 virtual visits at University Hospital Southampton.

It is safe to exercise and possible benefits include improved symptoms and quality of life. After exercising some people may feel achy or sore, but this should subside within a day or two. It is normal to feel short of breath during exercise. Occasionally, asthma symptoms are exacerbated briefly during exercise-this will be monitored for during the early supervised exercise sessions, and participants will be advised to take a dose of their reliever if needed.

During blood sampling, participants may feel discomfort due to the needle and may have bruising, bleeding or swelling at the blood sample site. Participants may feel faint and dizzy while blood is being drawn and there is a slight risk of infection.

Sometimes conversations about habits or emotional wellbeing might be a bit emotional but the Health Guide will be trained in how to provide support should this happen and to discuss further steps with participants if and when it is needed.

The study will open in the autumn of 2024, and will run for 18 months, with participants followed up for 12 months. The BMA James Trust is funding the study, with additional support from the NIHR

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 80 years Able and willing to give informed consent Diagnosis of asthma determined by

1. clinical diagnosis of difficult asthma as defined by BTS steps 4-5 and
2. enrolled in WATCH or meet WATCH inclusion criteria.
3. Demonstration of suboptimal symptom control through an ACQ ≥ 1.5 at enrolment
4. Normal lung function or mild/moderate airflow obstruction at baseline (FEV1>50% predicted)
5. Not achieving WHO recommendations for physical activity for people living with chronic health conditions(62) (150-300 minutes of moderate-intensity aerobic physical activity; or at least 75-150 minutes of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week) 6)12 lead ECG without clinically significant abnormality -

Exclusion Criteria:

1. Intercurrent exacerbation or exacerbation within 4 weeks prior to enrolment in study requiring treatment with oral corticosteroids and/or antibiotics. Note participants can be rescreened 4 weeks post exacerbation if they had not commenced the study
2. Initiation of biologic treatment within 6 months prior to recruitment or during study participation
3. Investigator determined significant change in regular asthma medication in the 12 weeks preceding or during trial period
4. Other medical or psychiatric conditions (including cognitive decline) limiting ability to exercise or that may in the opinion of the study clinician carry inherent risk for exercise
5. Contraindication to ISWT
6. Positive pregnancy test
7. Beta blocker treatment (due to impact on exercise prescription using HR) -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in Asthma Control Questionnaire score | pre and post intervention, at 12 month follow up
  Primary feasibility outcome is feasibility and acceptability to patients. Primary clinical endpoint outcome measure will be a minimal clinically significant improvement in ACQ 6 score (>0.5). Score scale is from 0-6, with < 1.5 demonstrating good asthma symptom control.

SECONDARY OUTCOMES:
Improvement in exercise capacity, QoL scores, exacerbation frequency | pre and post intervention, at 12 month follow up
  Increase in exercise capacity as assessed through oxygen uptake of > 2ml/kg/min at anaerobic threshold (AT) on maximal, symptom limited, incremental shuttle walk test.
Asthma Quality of Life Questionnaire (AQLQ) | pre and post intervention, at 12 month follow up
  32 questions scored on Likert scale 1-7. Score is mean of 32 answers, range 1-7 (higher =better quality of life
Exacerbation frequency | pre and post intervention, at 12 month follow up
  number of asthma exacerbations requiring oral corticosteroid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anna Freeman, MBBS PhD, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: No